CLINICAL TRIAL: NCT02007252
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Dose Study of Subcutaneous ACZ885 for the Treatment of Abdominal Aortic Aneurysm
Brief Title: ACZ885 for the Treatment of Abdominal Aortic Aneurysm
Acronym: AAA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The results of a third interim analysis (ad hoc) indicated a lack of efficacy and futility in continuing the trial.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CACZ885X2201; 2013-002088-25 (EudraCT Number)
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Results first posted 2016-11-21 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2019-03

CONDITIONS: Abdominal Aortic Aneurysm (AAA)
Keywords: Abdominal Aortic Aneurysm; AAA; IL-1b; Abdominal ultrasound
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACZ885 (Experimental): Participants received ACZ885 150 mg subcutaneously (s.c.) once per month for 12 months.
  Interventions: Drug: ACZ885
- Placebo (Placebo Comparator): Participants received matching placebo to ACZ885 s.c. once per month for 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACZ885 — ACZ885 150 mg liquid pre-filled syringes were administered s.c..
  Arms: ACZ885
Drug: Placebo — Matching placebo liquid pre-filled syringes were administered s.c..
  Arms: Placebo

SUMMARY:
This study was designed to assess the safety, tolerability and efficacy of ACZ885 on aneurysmal growth rate in subjects with abdominal aortic aneurysms (AAA). The purpose of the study was to provide data to enable decisions regarding the further development of ACZ885 for subjects with abdominal aortic aneurysms. The design of this study addressed the primary objective of evaluating the change in aneurysmal size in subjects with AAA as a result of treatment with ACZ885.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male and female subjects age ≥45 years of age
2. Infrarenal abdominal aortic aneurysm with maximum diameter: for men ≥40mm and ≤50mm; for women ≥38mm and ≤48mm.
3. On a stable medical regimen for at least 2 weeks prior to dosing, per investigator assessment.
4. Have an evaluable ultrasound image at screening for the quantitative determination of the AAA size, per imaging core lab assessment.
5. At screening, vital signs should be within the following ranges: (a) oral body temperature between 35.0-37.5°C; (b) systolic blood pressure, 90-170 mm Hg; (c) diastolic blood pressure, 50-100 mm Hg; (d) pulse rate, 40 - 100 bpm.

Key Exclusion Criteria:

1. Use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment.
2. Known diabetes by medical history, an HbA1c of ≥6.5% at screening, or on an active diabetic medical regimen.
3. History of malignancy of any organ system other than localized basal cell carcinoma of the skin, treated or untreated, within the past 5 years.
4. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during dosing and 30-day follow up period of the study.
5. Donation or loss of 400 ml or more of blood within eight (8) weeks prior to initial dosing, or longer if required by local regulation.
6. Subjects on the following medications: (a) Chronic systemic steroid treatment or other systemic immunosuppression; (b) Any biologic drugs targeting the immune system, along with a history of any previous use of such drugs.
7. Presence of a non-healing wound or infection, including active urinary tract infections, or any recent process requiring significant tissue healing per investigator assessment.
8. Significant illness which has not resolved within four (4) weeks prior to initial dosing or with a life expectancy less than 2 years.
9. Any of the following concomitant hepatic or renal conditions or diseases: (a) Nephrotic syndrome, or eGFR less than 30 mL/min/1.73 m2 per CRCL formula; (b) Prior organ transplant requiring immunosuppressive therapy; (c) Known active or recurrent hepatic disorder.
10. Previous infra-renal aortic surgery
11. Planned major surgery
12. Known aortic dissection
13. Subjects with eligible AAA diameter, but with known slow growth (<2mm/year) or known stable AAA size over the prior one year of surveillance per investigator assessment.
14. Subjects should exhibit no signs of clinically concerning unstable acceleration of AAA size or growth rate at the time of enrollment per investigator assessment.
15. Known or suspected inherited connective tissue disorders (e.g., Marfan or Vascular Ehlers Danlos syndrome).
16. Recently unstable clinically significant cardiac disease within 3 months of screening, including but not limited to, unstable angina, acute myocardial infarction, and congestive heart failure (NYHA class IV).
17. Uncontrolled or refractory hypertension per Investigator determination.
18. Live vaccinations within 3 months prior to randomization, or live vaccinations planned during the study.
19. History of untreated tuberculosis infection or evidence of active tuberculosis (TB) infection.
20. History of multiple and recurring allergies or allergy to the investigational compound/compound class being used in this study.
21. History of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result.
22. A positive Hepatitis B surface antigen or Hepatitis C test result whether at screening or historically.
23. For USA sites utilizing CT angiograms, subjects with a history of a previous reaction to contrast agent, a known sensitivity to iodine and known allergies (e.g, shellfish allergy), or other hypersensitivities to contrast agents.
24. Underlying immune disorders, autoimmunity or immunodeficiency.
25. History of drug or alcohol abuse within the 12 months prior to dosing.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Novartis Investigative Site, Charlottesville, Virginia, United States
- Denmark (3):
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Kolding
  - Novartis Investigative Site, Odense C
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Eindhoven
- Sweden (2):
  - Novartis Investigative Site, Örebro
  - Novartis Investigative Site, Stockholm
- Novartis Investigative Site, Manchester, United Kingdom

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=81

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 65 participants were randomized in a 1:1 ratio to one of the two treatment groups. One participant discontinued prior to taking any study medication. As such, the participant flow is based on 64 randomized participants.
Period: Overall Study
Arm/Group | ACZ885 | Placebo
Started | 31 | 33
Safety Analysis Set | 31 | 33
Pharmacodynamic Analysis Set | 31 | 33
Completed | 20 | 22
Not Completed | 11 | 11
Not completed — Administrative problems | 3 | 7
Not completed — Abnormal laboratory value(s) | 1 | 0
Not completed — Adverse Event | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACZ885 | Placebo | Total
Number analyzed (Participants) | 31 | 33 | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.4 (7.44) | 70.8 (5.84) | 70.1 (6.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 27 | 26 | 53

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Abdominal Aortic Aneurysm (AAA) Size Per Year
Description: Size of the AAA was determined using an abdominal ultrasound technique at baseline, 3 months, and 12 months after treatment with study drug. Growth rate (in mm/year) was calculated from the change in AAA size compared to baseline
Time Frame: month 3, month 12
Population: The pharmacodynamic analysis set, which included randomized participants who received at least one dose of study drug, was considered for the analysis. However, only participants with values at each time point were analyzed.
Measure: Least Squares Mean (90% Confidence Interval); unit: millimeter/year
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 31 | 33
millimeter/year
  Month 3 (n=23,31) | 0.781 [-0.942 to 5.504] | 2.519 [1.030 to 4.008]
  Month 12 (n=20,23) | 2.538 [1.465 to 3.612] | 2.581 [1.612 to 3.549]
Statistical Analysis 1: Comparison: ACZ885 vs Placebo; Month 3; Test type: Superiority or Other; p = 0.1037, ANCOVA
Statistical Analysis 2: Comparison: ACZ885 vs Placebo; Month 12; Test type: Superiority or Other; p = 0.4806, ANCOVA

ADVERSE EVENTS:
Arm/Group | ACZ885 | Placebo
Serious Adverse Events (participants affected / at risk) | 2/31 | 0/33
Other Adverse Events (participants affected / at risk) | 28/31 | 28/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACZ885 (N=31) | Placebo (N=33)
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACZ885 (N=31) | Placebo (N=33)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Energy increased (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
Impaired healing (General disorders) | 1 | 1
Influenza like illness (General disorders) | 0 | 1
Injection site hypersensitivity (General disorders) | 1 | 0
Injection site pain (General disorders) | 1 | 1
Injection site swelling (General disorders) | 3 | 2
Malaise (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 4
Erysipelas (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 5 | 3
Pneumonia (Infections and infestations) | 2 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 2 | 1
Vestibular neuronitis (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2
Blood creatinine increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0
Occult blood positive (Investigations) | 2 | 0
Prostatic specific antigen increased (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 0
Sciatica (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1
Breast cyst (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 2
Hot flush (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 4 | 3
Intermittent claudication (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.